CLINICAL TRIAL: NCT05312606
Title: Domiciliary Use of Hyaluronic Acid Gel Solutions vs Domiciliary Use of Chlorhexidine Mouthwash 0,20% for the Management of Periodontal Patients: a Randomized Clinical Trial
Brief Title: Domiciliary Use of Hyaluronic Acid Gel Solutions vs Domiciliary Use of Chlorhexidine Mouthwash 0,20% for the Management of Periodontal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-AFTORAL PARO
Record Dates: First submitted 2022-03-26; First posted 2022-04-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Home treatment with hyaluronic acid.
  Interventions: Other: Aftoral Oral gel
- Control Group (Active Comparator): Home treatment with chlorhexidine.
  Interventions: Other: Unidea Chlorhexidine digluconate mouthwash 0.20%

INTERVENTIONS:
Other: Aftoral Oral gel — Patients will use Aftoral® Oral Gel solution for the domiciliary application once a day for 15 days after the visits (no rinsing and eating for 30 minutes after gel solution application).
  Arms: Trial Group
Other: Unidea Chlorhexidine digluconate mouthwash 0.20% — Patients will use chlorhexidine mouthwash 0,20% for the domiciliary application once a day for 15 days after the visits (no rinsing and eating for 30 minutes after mouthwash application).
  Arms: Control Group

SUMMARY:
Brief Summary: This is a randomized controlled clinical trial (RCT). After signing the informed consent, patients satisfying the inclusion criteria will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation, manual instrumentation with Gracey curettes and air polishing with glycine powder.

After that, the sample will be randomly divided into 2 groups based on the domiciliary assigned treatment:

* Aftoral® Oral Gel solution with Hyaluronic Acid, Xylitol and glycerophosphoinositol as a domiciliary application for 15 days.
* Unidea® Chlorhexidine digluconate Mouthwash 0,20% administration as a domiciliary application for 15 days.

The study will last 6 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), after 6 months (T3). Professional hygiene will be performed again at T2 and T3.

At each recall session were collected a satisfaction questionnaire of the products (taste, smell, consistency, persistence and ease of application) and the following periodontal clinical indices, using a Periodontal probe on each site:

* Gingival Recession (R)
* PPD (Probing Pocket Depth),
* BOP% (Bleeding on Probing),
* CAL (Clinical Attachment Level),
* PCR% (Plaque Control Record),
* Tooth Mobility.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial (RCT). 40 patients are expected to be enrolled. After signing the informed consent, patients satisfying the inclusion criteria will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation, manual instrumentation with Gracey curettes and air polishing with glycine powder.

All patients will be treated at the Unit of Dental Hygiene, Section of Dentistry, Department of Clinical, Surgical, Diagnostic, and Pediatric Sciences of the University of Pavia.

After that, the sample will be randomly divided into 2 groups based on the domiciliary assigned treatment:

* Aftoral® Oral Gel solution with Hyaluronic Acid, Xylitol and glycerophosphoinositol as a domiciliary application for 15 days.
* Unidea® Chlorhexidine digluconate Mouthwash 0,20% administration as a domiciliary application for 15 days.

The study will last 6 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), and after 6 months (T3).

At T2 and T3, professional hygiene will be performed again.

At each recall session were collected a satisfaction questionnaire of the products (taste, smell, consistency, persistence and ease of application) and the following periodontal clinical indices, using a Periodontal probe on each site:

* Gingival Recession (R),
* PPD (Probing Pocket Depth),
* BOP% (Bleeding on Probing),
* CAL (Clinical Attachment Level),
* PCR% (Plaque Control Record),
* Tooth Mobility.

ELIGIBILITY:
Inclusion Criteria:

* presence of stage II periodontitis sistes according to the 2017 World Workshop classification system
* no systemic, metabolic and autoimmune disease
* compliant patients

Exclusion Criteria:

* neurologic, psychiatric and mental diseases
* patients taking bisphosphonates in the last 12 months
* patients taking antibiotics during the study
* pregnant and breastfeeding women
* patients undergoing anticancer treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Gingival Recession (R) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Evaluation (in mm) of the displacement of marginal tissue, through a millimeter periodontal probe; it is detected from the cemento-enamel junction (CEJ) to the gingival margin.
Change in Bleeding on Probing (BOP%) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Quantitative assessment (percentage) of the bleeding sites (6 per tooth in total).
  Formula = n ° bleeding sites / n ° probed sites x100
Change in Clinical Attachment Level (CAL) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Evaluation (in mm) of the distance of the cemento-enamel junction (CEJ) to the bottom of the gingival sulcus or periodontal pocket, evaluated in 6 sites.
Change in Plaque Control Record (PCR%) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
  Formula = n ° sites with plaque / total n ° of dental surfaces x100

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data are available upon motivated request to the Principal Investigator.